CLINICAL TRIAL: NCT05468567
Title: Three-dimensional Perception of Sounds in Military with Acoustic Trauma
Acronym: SPHEAR
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0692
Record Dates: First submitted 2022-07-01; First posted 2022-07-21 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Hearing Loss
Keywords: Spatial hearing; virtual reality; acoustic trauma; hearing loss
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Noise-Induced

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Military person with acoustic trauma (experimental group): Active or reserve military member, diagnosed with acoustic trauma for at least one month. Participants will be instructed to localize a sound emitted in their environment using a virtual reality setup.
  Interventions: Diagnostic Test: SPHERE protocol : Spatial hearing performances test; Diagnostic Test: French Matrix Test : audiology test of speech in noise perception; Behavioral: SSQ15 questionnaire of life : (The Speech, Spatial and Other Qualities of Hearing Scale)
- Normal hearing volunteers (control group): Person without known hearing loss.
  Interventions: Diagnostic Test: SPHERE protocol : Spatial hearing performances test; Diagnostic Test: French Matrix Test : audiology test of speech in noise perception; Behavioral: SSQ15 questionnaire of life : (The Speech, Spatial and Other Qualities of Hearing Scale)

INTERVENTIONS:
Diagnostic Test: SPHERE protocol : Spatial hearing performances test — Participants will be instructed to localize a sound emitted in their environment using a virtual reality setup (SPHEAR protocol).
Diagnostic Test: French Matrix Test : audiology test of speech in noise perception — Intelligibility threshold is the signal-to-noise ratio (in decibels) for which the subject can repeat 50% of the words heard in a dichotic listening.
Behavioral: SSQ15 questionnaire of life : (The Speech, Spatial and Other Qualities of Hearing Scale) — The SSQ questionnaire is a clinical subjective scale that allows evaluating of hearing performances in daily life. The questionnaire is divided into 3 main items (A: speech; B: spatial hearing; C: other qualities of hearing) comprising questions with rating scores out of ten.

SUMMARY:
Spatial hearing capacities of soldiers with acoustic trauma are evaluated in ENT consultations with routine tests (i.e. tonal audiometry, voice audiometry). While the results conclude that soldiers with acoustic trauma have sufficient abilities to carry out professional missions, soldiers report recurring complaints of sound localization (spatial hearing), i.e. difficulties in identifying the position of sound sources in their environment. However, there is currently no objective test to identify and objectify these complaints of spatial hearing.

The investigators have developed a new approach (SPHERE) based on virtual reality and 3D motion tracking, allowing us to evaluate and record the spatial hearing performance of subject with hearing deficit. This system allowed us to highlight localization deficits in three-dimensional space.

This project explores and quantifies the spatial hearing impairments of soldiers with acoustic trauma. The quantification of the spatial hearing capacities will allow to define a specific rehabilitation strategy of spatial hearing deficits.

ELIGIBILITY:
Inclusion Criteria:

acoustic traumatized military group :

* Age between 18 and 65 inclusive
* Active or reserve military personnel
* Diagnosis of noise trauma for at least one month
* Regularly followed up in the ENT department of the Desgenettes Army Training Hospital in Lyon or in the medical offices of the Army Medical Centers.
* Able to understand the experimental instructions
* Affiliated to a social security scheme
* Having been informed of the study and having given their agreement to participate normal hearing group :
* Age between 18 and 65 years inclusive
* Able to understand the experimental instructions
* Affiliated to a social security scheme
* Having been informed of the study and given their agreement to participate

Exclusion Criteria:

* Known current or past neurological or psychiatric disorder
* Oculomotor/visual disorder
* Bilateral vestibular areflexia
* Person under court protection, guardianship or curatorship
* Pregnant or breastfeeding woman
* Known hearing loss for normal hearing group

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Army Training Hospital of Lyon or within the medical branches of the Army Medical Centers are the structures where the soldiers will recruited. The Neurosciences research Center of Lyon or the ENT department of Edouard Herriot Hospital will recruit the normal hearing volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative error value "3d-D" measuring the spatial hearing performances | at Day 1 during the inclusion visit. The test last 30 minutes.
  First, the pointing error will be computed for azimuth, elevation, and depth, in terms of constant error and variable error. Then, these separate dimension errors will be combined into a cumulative error "3d-D", taking into account absolute and variable error in one measure. 3d-D value corresponding to the spatial hearing deficit matching the distance between the 3D hand pointing position and the 3D sound source position.
  The 3dD performance of the Acoustic traumatised military group will be compared to that of the normal hearing group.

SECONDARY OUTCOMES:
Correlation between the score obtained in the SSQ and the 3dD auditory spatialization performance. | at Day 1 during the inclusion visit.
  The behavioral (dependent) variables from the SSQ of the acoustic traumatized military will be analyzed using the linear regression method to examine the relationship between their 3dD auditory spatialization performance and their SSQ score
Correlation between the score obtained in the Framatrix and the 3dD auditory spatialization performance. | at Day 1 during the inclusion visit.
  The speech-in-noise performance (SNR) of the acoustic traumatized military will be analysed using the linear regression method to examine the relationship between their speech-in-noise performance (SNR) and their SSQ score

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Edouard Herriot, Lyon, France